CLINICAL TRIAL: NCT01154972
Title: Preoperative Identification of the Sentinel Lymph Node in Breast Cancer, Using Ultrasound and Radio-isotope/Percutaneous Gamma Probe
Brief Title: Preoperative Localisation of the Sentinel Lymph Node in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Tayside (Other Government)
Collaborators: University of Dundee (Other)
Responsible Party: Principal Investigator, Andy Evans, Professor of Breast Imaging, NHS Tayside
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010ON03
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer
Keywords: breast; cancer; sentinel lymph node
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm study - Sentinel Node Localisation (Experimental)
  Interventions: Procedure: Preoperative sentinel lymph node identification and marking

INTERVENTIONS:
Procedure: Preoperative sentinel lymph node identification and marking — SLN is identified using gamma probe and ultrasound. Percutaneous wire placement carried out to mark SLN for subsequent surgical verification.

SUMMARY:
When a person has breast cancer it is necessary to find out whether the cancer has spread to the lymph nodes in the armpit because if it has, further treatment is likely to be needed. There are many of these nodes but when the breast cancer spreads, it does so in a step-by-step fashion, starting with the so-called Sentinel Lymph Node (SLN). At present, the only way to be sure whether there is cancer in the lymph nodes or not is to perform an operation to remove at least the SLN. If the pathologist finds cancer in the SLN, a second operation is usually required to remove further nodes in case they contain cancer too. Surgical removal of the lymph nodes in the armpit can cause difficulties for the patient afterwards, such as pain and swelling in the arm. If there is no cancer in the SLN, no further operations on the armpit are needed. The investigators wish to find out whether in some patients, operations on the armpit can be avoided completely. The first step in doing this is to test whether the investigators can find out which is the SLN before the operation, using a combination of an injection and ultrasound scanning. The injection - into the skin of the breast - would be a radioactive substance, which is the usual way the surgeon finds the SLN. The radioactive substance collects in the SLN and the investigators would use a "gamma probe" over the surface of the armpit to detect the radiation. In this initial study, the investigators would aim to find the SLN before the operation and place a marker wire in it so that the surgeon could check whether the investigators had found the correct node.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with invasive breast cancer suitable for primary surgical treatment
* Booked for surgical Sentinel Lymph Node Biopsy

Exclusion Criteria:

* Unable to give informed consent
* Known bleeding disorder
* Previous axillary surgery
* Previously treated for the current tumour with chemotherapy or hormone therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-04; Primary Completion 2012-11-01 (Actual); Study Completion 2013-05-10 (Actual)

PRIMARY OUTCOMES:
Is the sentinel lymph node marked preoperatively confirmed as the SLN at surgery? | 8 Months from start of trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Ninewells Hospital and Medical School, Dundee, United Kingdom